CLINICAL TRIAL: NCT04856657
Title: Targeting Individual Alpha Frequencies to Enhance Perceptual Timing
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: PSYCH-2021-29530
Record Dates: First submitted 2021-04-13; First posted 2021-04-23 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Psychosis; Schizophrenia; Schizo Affective Disorder
Keywords: tacs; neuromodulation; psychosis; schizophrenia
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Spondylocostal Dysostosis 4, Autosomal Dominant | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Session 1: tACS at IAPF + 2 Hz: Participants in this arm will undergo tACS at a frequency 2 Hz above their IAPF during stimulation session 1. They will undergo tACS at a frequency 2 Hz below their IAPF during stimulation session 2.
  Interventions: Device: Transcranial alternating current stimulation
- Session 1: tACS at IAPF - 2 Hz: Participants in this arm will undergo tACS at a frequency 2 Hz below their IAPF during stimulation session 1. They will undergo tACS at a frequency 2 Hz above their IAPF during stimulation session 2.
  Interventions: Device: Transcranial alternating current stimulation

INTERVENTIONS:
Device: Transcranial alternating current stimulation — The tACS will be applied with a current of 1-2 mA (milliamperes) via two saline soaked electrode sponges (25 cm²) applied to the back of the head. The anode will be located at Oz and the cathode will be located at Cz.
  Other Names: tACS

SUMMARY:
This is a single-blind randomized within-subject crossover design study that will be conducted in 2 phases. In Phase 1, up to 50 participants, after signing informed consent and determining eligibility, will undergo a baseline EEG and cognitive assessment. In Phase 2 participants will undergo tACS at IAF+2Hz, IAF-2Hz, and IAF during a double-flash illusion task in a randomized order. The tACS will be applied with a current of 1-2 mA (milliamperes) via two saline soaked electrode sponges (25 cm²) applied to the back of the head. The investigator's hypothesis is that participant's will perform better on the visual task while tACS is set to 2 Hz above their IAPF, relative to tACS set to 2 Hz below their IAPF.

DETAILED DESCRIPTION:
The proposed pilot study will assess the feasibility of transcranial alternating current stimulation (tACS) to enhance aspects of attention in people with psychotic disorders.

If a participant agrees to participate in this research, they will be asked to visit the study site to complete the activities listed below. These study activities will take about 5.5 hours to complete. The activities can be divided into up to 3 separate sessions as needed, but all activities should be completed within approximately one week.

Phase 1:

* A clinical interview including an abbreviated MINI, consisting of the mood, mania, suicide, and psychosis modules to either: confirm a diagnosis of a psychotic disorder in Psychosis Subject recruits; or confirm no diagnosis of a psychotic disorder in Control Subject recruits. If any suicidal ideation is expressed on the suicide module, study staff will administer the C-SSRS.
* All participants will complete the Wechsler Test of Adult Reading (WTAR) to obtain an estimate of average IQ, the Brief Assessment of Cognition (BAC app; including Verbal Learning, Digit Sequencing, Token Motor, Semantic Fluency, Symbol Coding, and Tower of London), the Edinburgh Handedness Inventory, and a brief demographic questionnaire.
* Participants with psychosis will complete the PANSS clinical interview to assess psychosis symptoms. Controls will not complete the PANSS.
* Next, participants will undergo a baseline EEG that includes measures of resting EEG (once at the beginning and once more at the end of the session) and a Double-Flash Fusion Illusion Task.

Phase 2:

* Participants will undergo a shortened version of the Double-Flash task without any tACS stimulation.
* Participants will then undergo 3 shortened versions of the Double-Flash Fusion Illusion task while simultaneously undergoing tACS. In counterbalanced order, participants will have tACS set at their IAF (obtained from the subject's resting EEG signal), their IAF + 2Hz and their IAF - 2 Hz. Each task run is expected to last 10-20 minutes. In the first ~1 minute of stimulation before starting the task, we will ask participants to report whether they are perceiving phosphenes. We will turn down the stimulation in .1 mA increments until the participant is no longer perceiving bothersome phosphenes before starting the task. Participants will have a ~40 minute break between task sessions.
* During one of the 40 minute between session breaks, participants will be asked to perform two assessment versions of a time-order frequency judgment task: Sound Sweeps (auditory frequency modulation time-order judgement) and Visual Sweeps (visual gabor frequency modulation time-order judgement).
* Following the third stimulation/task session, participants will respond to a questionnaire about the tolerability of the stimulation and whether they experienced any immediate adverse effects.

  * Currently, subjects will only undergo Phase 1 of the study to optimally pilot test the task and EEG procedures prior to enrolling subjects to both Phases which involves an experimental manipulation of the Double-Flash task. Phase 2 will be initiated at the discretion of the PI.

ELIGIBILITY:
Psychosis Participants:

Inclusion Criteria:

* Meet diagnostic criteria for a psychotic disorder (schizophrenia, schizoaffective disorder, schizophreniform disorder, major depressive disorder with psychotic features, bipolar disorder with psychotic features, psychosis disorder not otherwise specified, or unspecified schizophrenia spectrum disorder), as defined by the MINI (Mini-International Neuropsychiatric Interview)
* Are age 18-64 (inclusive)
* Fluent in written and spoken English
* Have an outpatient status of at least 1 month prior to participation
* Has been on a stable dose of psychiatric medication for at least one month prior to participation (titration to a lower dose of psychotropic medications under supervision of a psychiatrist can be allowed at the discretion of the investigators)

Exclusion Criteria:

* History of seizures or epilepsy
* Metallic cranial plates, screws, or implanted devices
* History of craniotomy
* History of stroke
* History of eczema on scalp
* Pre-existing sores or lesions at sites of tACS electrode placement
* Non-removable facial piercings
* Current or possibility of current pregnancy
* Active suicidal ideation at screening or baseline assessments, or previous intent to act on suicidal ideation with a specific plan, preparatory acts, or an actual suicide attempt within the last 3 months, as indicated by the MINI and/or C-SSRS (All participants will complete the suicide module of the MINI. If participants express any suicidal ideation on the MINI, staff will complete the C-SSRS [Columbia-Suicide Severity Rating Scale].)
* WTAR (Wechsler Test of Adult Reading) standardized score below 70
* Any reason our tCS (transcranial stimulation) or EEG caps cannot be placed on their head

Control Participants:

Inclusion Criteria:

* Are age 18-64 (inclusive)
* Fluent in written and spoken English

Exclusion Criteria:

* Meet diagnostic criteria for a psychotic disorder (schizophrenia, schizoaffective disorder, schizophreniform disorder, major depressive disorder with psychotic features, bipolar disorder with psychotic features, psychosis disorder not otherwise specified, or unspecified schizophrenia spectrum disorder), as defined by the MINI
* Self-reports having a first-degree relative with a psychotic disorder
* History of seizures or epilepsy
* Metallic cranial plates, screws, or implanted devices
* History of craniotomy
* History of stroke
* History of eczema on scalp
* Pre-existing sores or lesions at sites of tACS electrode placement
* Non-removable facial piercings
* Current or possibility of current pregnancy
* Active suicidal ideation at screening or baseline assessments, or previous intent to act on suicidal ideation with a specific plan, preparatory acts, or an actual suicide attempt within the last 3 months, as indicated by the MINI and/or C-SSRS (All participants will complete the suicide module of the MINI. If participants express any suicidal ideation on the MINI, staff will complete the C-SSRS.)
* WTAR standardized score below 70
* Any reason our tCS or EEG caps cannot be placed on their head

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study will study individuals who experience psychosis, including schizophrenia, schizoaffective disorder, and bipolar disorder with psychosis.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2023-02-09 (Actual)

PRIMARY OUTCOMES:
Double Flash Fusion Illusion Task | 2 20-minute task runs (one during tACS at IAPF + 2 Hz and one during tACS at IAPF - 2 Hz)
  Participants are instructed to fixate their gaze on a central fixation cross. When the cue appears, a low-luminance disc stimulus flashes on either side (left or right) of the fixation cross. The disc can flash one or two times. After the stimulus ends, participants are cued to make a response regarding the number of disc flashes (1 or 2). Participants will undergo 300 trials. Participants will be scored on response accuracy (i.e., number of correct responses out of 300 possible responses).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States